CLINICAL TRIAL: NCT07169565
Title: Phase I Clinical Study of Ibrutinib Followed by BR (Bendamustine and Rituximab) as a Time-Limited Therapy for Waldenström Macroglobulinemia
Brief Title: Ibrutinib Followed by BR (Bendamustine and Rituximab) as a Time-Limited Therapy for Waldenström Macroglobulinemia
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2022026
Record Dates: First submitted 2025-07-31; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Waldenström Macroglobulinemia (WM)
Keywords: Waldenström Macroglobulinemia; ibrutinib; fixed dose
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — ibrutinib; Bendamustine Hydrochloride; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Ibrutinib + BR Combination Therapy (Experimental): 1. A 3+3 dose-escalation phase to determine the Maximum Tolerated Dose (MTD) and Recommended Phase II Dose (RP2D) of the I+BR regimen in Waldenström Macroglobulinemia (WM) patients;
  2. A dose-expansion phase to evaluate the safety, tolerability, and efficacy of the time-limited regimen at the MTD/RP2D.
  Interventions: Drug: Ibrutinib; Drug: Bendamustine; Drug: Rituximab

INTERVENTIONS:
Drug: Ibrutinib — Oral Bruton's tyrosine kinase (BTK) inhibitor administered at a fixed dose of 420 mg once daily. Capsules must be swallowed whole with water; do not open, break, or chew. If a dose is missed by ≤6 hours, take immediately; if >6 hours, skip the dose and resume normal schedule the next day. Avoid grapefruit and Seville oranges (moderate CYP3A inhibitors). Treatment duration: 3 cycles (28 days/cycle) or until disease progression/unacceptable toxicity. Dose reduction is mandated for specific toxicities: 420 mg → 280 mg → 140 mg → discontinuation (per protocol-specified criteria). Use with caution in hepatic impairment (Child-Pugh A: reduce to 80 mg/day; Child-Pugh B/C: contraindicated).
Drug: Bendamustine — Intravenous alkylating agent dosed via a 3+3 dose de-escalation design (70 mg/m² → 60 mg/m² → 50 mg/m²). Infused over 60-120 minutes on Days 1-2 of each 28-day cycle for 3 cycles. Starting dose: 70 mg/m² (Dose Level 1); dose reduction triggered by Dose-Limiting Toxicity (DLT) events per protocol. In the dose-expansion phase, all subjects receive the MTD/RP2D established in Part 1. Concomitant live vaccines are prohibited. Dose delays (≤4 weeks) and reductions are required for Grade ≥3 hematologic/non-hematologic toxicities.
Drug: Rituximab — Intravenous anti-CD20 monoclonal antibody administered at a fixed dose of 375 mg/m² on Day 0 of each 28-day cycle for 3 cycles. Initial infusion starts at 50 mg/hour; if tolerated, increase by 50 mg/hour every 30 minutes (maximum: 400 mg/hour). Subsequent infusions start at 100 mg/hour with the same escalation. Premedication with acetaminophen and an antihistamine is required prior to each infusion. Permanently discontinue for Grade 4 infusion-related reactions or severe/life-threatening toxicity.

SUMMARY:
This is a two-part, non-randomized, open-label Phase I clinical study. The research consists of:

1. A 3+3 dose-escalation phase to determine the Maximum Tolerated Dose (MTD) and Recommended Phase II Dose (RP2D) of the I+BR regimen in Waldenström Macroglobulinemia (WM) patients;
2. A dose-expansion phase to evaluate the safety, tolerability, and efficacy of the time-limited regimen at the MTD/RP2D.

Key Study Design Details:

Pre-enrollment & Eligibility:

* Patients undergo efficacy and tolerability assessment before enrollment.
* Eligible patients receive I+BR therapy.

Treatment Regimen:

* Bendamustine: Tested at three dose levels (70 mg/m², 60 mg/m², and 50 mg/m²) based on prior IBR data in B-cell lymphomas. A 3+3 dose de-escalation design is employed.
* Fixed Doses:

  * Ibrutinib: 420 mg/day
  * Rituximab: 375 mg/m²

Part I (3+3 Dose Escalation):

* Start with 3 patients receiving bendamustine 70 mg/m².
* After 1 treatment cycle:

  * Assess Dose-Limiting Toxicity (DLT) (DLT criteria defined separately).
  * Patients without DLT proceed to 2 additional cycles of IBR.
* After 3 total cycles:

  * Efficacy assessment is performed.
  * Patients achieving minimal response (MR) or better (i.e., MR, PR, VGPR, CR) receive 1 cycle of BR, then cease treatment and enter follow-up.
  * Patients failing to achieve ≥MR are withdrawn.
* Primary Objective: Evaluate safety and identify MTD.

Part II (Dose Expansion):

* Enroll 15 additional patients at MTD/RP2D.
* Objectives:

  * Further assess safety and efficacy;
  * Monitor IgM rebound within 2 months after completing therapy (3 cycles I+BR → 1 cycle BR);
  * Explore correlations between biomarkers and clinical outcomes.

Terminology Notes:

* I+BR: Ibrutinib + Bendamustine/Rituximab
* DLT: Dose-Limiting Toxicity
* MTD: Maximum Tolerated Dose
* RP2D: Recommended Phase II Dose
* Efficacy thresholds: MR (Minimal Response), PR (Partial Response), VGPR (Very Good Partial Response), CR (Complete Response)
* Time-limited therapy: Fixed-duration treatment designed to avoid indefinite dosing.

ELIGIBILITY:
Inclusion Criteria

1. Patient fully understands the study, voluntarily participates, and signs the Informed Consent Form (ICF).
2. Patient of any gender, aged ≥18 years and ≤75 years.
3. Patient must meet diagnostic criteria for Waldenström Macroglobulinemia (WM) and be MYD88 L265P mutation positive.
4. Patient has documented baseline IgM levels and disease assessment parameters (including liver, spleen, lymph nodes; if extramedullary lesions exist, include assessment of other extramedullary sites) prior to ibrutinib use, to facilitate subsequent efficacy evaluation.
5. ECOG performance status score of 0-1.
6. Patient has received ≥12 cycles of ibrutinib monotherapy, achieved a treatment response (but not Complete Response (CR) ), and is currently on a treatment plateau.
7. Patient has maintained good treatment tolerance (experienced no Grade ≥3 adverse reactions during ibrutinib therapy) and is still receiving ibrutinib.
8. Patient has no prior treatment with Bendamustine combined with Rituximab (BR) regimen.
9. Laboratory values:

   * Neutrophils ≥1.0 × 10⁹/L
   * Platelets ≥50 × 10⁹/L
   * Hemoglobin ≥70 g/L
   * Total bilirubin ≤2 × Upper Limit of Normal (ULN)
   * Alanine aminotransferase (ALT) / Aspartate aminotransferase (AST) ≤3 × ULN
   * Creatinine clearance (CrCl) ≥30 mL/min (calculated by Cockcroft-Gault formula).
10. Patient has an estimated life expectancy ≥6 months.

Exclusion Criteria

1. Diagnosis or treatment for a malignancy other than B-cell Non-Hodgkin Lymphoma (B-NHL) within the past year (including active Central Nervous System lymphoma). Received other anti-tumor therapies (including chemotherapy, targeted therapy, hormonal therapy, anti-tumor Chinese herbs with activity) within 4 weeks prior to study drug administration (excluding ibrutinib) or participated in other clinical trials receiving investigational drugs.
2. Clinical evidence of transformation to large cell lymphoma.
3. Non-lymphoma related liver or kidney impairment:

   * ALT >3 × ULN
   * AST >3 × ULN
   * Total bilirubin (TBIL) >2 × ULN
   * Serum creatinine clearance <30 mL/min.
4. Other severe medical conditions that could interfere with the study (e.g., uncontrolled diabetes, gastric ulcer, other severe cardiopulmonary diseases), as determined by the investigator.
5. Cardiac function or disease meeting any of the following:

   1. Long QTc syndrome or QTc interval >480 ms;
   2. Complete left bundle branch block, second- or third-degree atrioventricular block;
   3. Severe, uncontrolled arrhythmias requiring drug therapy;
   4. New York Heart Association (NYHA) classification ≥ Class III;
   5. Left ventricular ejection fraction (LVEF) <50%;
   6. History within 6 months prior to enrollment: myocardial infarction, unstable angina, severe unstable ventricular arrhythmias, or any other arrhythmia requiring treatment; history of clinically significant pericardial disease; or ECG evidence of acute ischemia or active conduction system abnormalities.
6. Known history of Human Immunodeficiency Virus (HIV) infection, or active Hepatitis B Virus (HBV) infection, or any uncontrolled active systemic infection requiring intravenous antibiotics.

   Note: Active HBV infection is defined as meeting ALL THREE criteria: a. HBV DNA quantification ≥2000 IU/mL; b. ALT ≥2 × ULN; c. Hepatitis not attributable to other causes (e.g., disease itself, drugs). Patients initially diagnosed with active HBV infection who convert to inactive HBV status after anti-HBV therapy may be enrolled provided they receive adequate anti-HBV prophylaxis.
7. Major surgery within 14 days prior to enrollment (excluding lymph node biopsy) or anticipated need for major surgery during the study.
8. History or current diagnosis of another malignancy (except adequately controlled non-melanoma skin basal cell carcinoma, carcinoma in situ of the breast/cervix, and other malignancies effectively controlled without treatment for the past five years).
9. Pregnant or lactating women, or women of childbearing potential not using contraception.
10. Hypersensitivity to any of the study drugs or their components.
11. Malabsorption syndrome, disease significantly affecting gastrointestinal function, gastrectomy, extensive small bowel resection potentially affecting absorption, symptomatic inflammatory bowel disease, partial or complete bowel obstruction, or gastric restriction/bariatric surgery (e.g., gastric bypass).
12. History of stroke or intracranial hemorrhage within 6 months prior to the first dose of study drug.
13. History of bleeding diathesis (e.g., hemophilia, von Willebrand disease).
14. Requirement for or ongoing anticoagulation therapy with warfarin or equivalent vitamin K antagonists (e.g., phenprocoumon) within 7 days prior to the first dose of study drug.
15. Diagnosis of gastrointestinal ulcer by endoscopy within 3 months prior to the first dose of study drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Dose Escalation (Part 1) Incidence of Dose-Limiting Toxicities (DLTs) | Cycle 1 (Days 1-28)
  Proportion of participants experiencing protocol-defined DLTs during Cycle 1 (28 days). DLTs include Grade ≥3 non-hematologic or specific hematologic toxicities (e.g., febrile neutropenia, Grade 4 thrombocytopenia >7 days) attributed to IBR regimen per NCI CTCAE v4.0 criteria (Section 2.4).
Phase 1: Dose Escalation (Part 1) Maximum Tolerated Dose (MTD) of Bendamustine | End of Dose Escalation Phase (approximately 6 months)
  Highest dose level (70/60/50 mg/m²) at which ≤1 of 6 participants experience DLTs during Cycle 1, determined via 3+3 dose-escalation design (Section 2.1).
Phase 1: Dose Escalation (Part 1) Recommended Phase 2 Dose (RP2D) | End of Dose Escalation Phase (approximately 6 months)
  Optimal dose of Bendamustine for expansion phase, derived from MTD evaluation integrated with safety/tolerability data (Section 2.1).
Phase 2: Dose Expansion (Part 2) Treatment-Emergent Adverse Events (TEAEs) at RP2D | From first dose until 30 days after last dose (up to 5 months)
  Frequency and severity of TEAEs (Grade ≥3 per NCI CTCAE v4.0) attributed to IBR regimen at the RP2D. Includes hematologic, non-hematologic, and serious adverse events.
Phase 2: Dose Expansion (Part 2) Overall Response Rate (ORR) at RP2D | At end of Cycle 3 (Day 84 ±3 days)
  Proportion of participants achieving ≥Partial Response (PR) per Consensus Panel Criteria from the 8th International Workshop on Waldenström Macroglobulinemia (IWWM-8) after 3 cycles of IBR therapy.

SECONDARY OUTCOMES:
IgM rebound rate | At 2 months after the last dose of study treatment
  Proportion of participants experiencing an IgM rebound, defined as a ≥25% increase in serum IgM levels from the end-of-treatment measurement, within 2 months after discontinuation of the time-limited therapy.
Duration of Response (DOR) | From the first documented response until disease progression/recurrence (assessed up to 24 months)
  Time from the date of initial documented response (partial response or better) to the date of documented disease progression or death from any cause, whichever occurs first.
Progression-Free Survival (PFS) | From first dose until disease progression or death (assessed up to 24 months)
  Time from the first dose of study drug to the date of documented disease progression or death from any cause, whichever occurs first.
Biomarker correlation with efficacy | Biomarker samples collected at baseline; efficacy assessed through study completion (approximately 24 months)
  Assessment of the association between specific biomarker levels (e.g., CXCR4 mutation status) and clinical efficacy outcomes (e.g., overall response rate).

OTHER OUTCOMES:
Correlation of Baseline Biomarker Status with Treatment Efficacy | Biomarker status: At screening (Day -28 to Day 1); Efficacy assessment: At the end of Cycle 3 (Day 84)
  To assess the association between the presence of specific somatic mutations (e.g., MYD88, CXCR4) detected at baseline and the achievement of a clinical response (Partial Response or better as defined by IWWM-8 criteria) following combination therapy. The strength of the association will be measured using odds ratios from logistic regression analysis.
Biomarker Correlation with Adverse Reactions | Biomarker samples collected at baseline (Day 1 Cycle 1); safety assessed from first dose until 30 days after last dose (approximately 24 months)
  To assess the impact of specific biomarkers (e.g., pharmacogenetic variants) on the incidence and severity of treatment-emergent adverse events (e.g., neutropenia, rash) after combination therapy. The association will be analyzed using appropriate statistical tests.
Temporal Changes in Biomarker Burden | Baseline (screening) vs. End of Cycle 3 (Day 84 ±3 days)
  Quantitative changes in mutation burden (e.g., MYD88 L265P variant allele frequency) from baseline to end of Cycle 3, measured by ddPCR in bone marrow/peripheral blood samples.
Impact of Germline Genetic Variants on Incidence of Specific Adverse Reactions | Genetic variant status: At screening (Day -28 to Day 1); Safety assessment: From first dose until 30 days after last dose (up to 24 weeks) Summary of Revisions:
  To evaluate the relationship between predefined germline pharmacogenetic variants (e.g., in genes encoding CYP metabolizing enzymes) and the occurrence of specific Grade ≥3 adverse events (e.g., neutropenia, rash) attributed to the study regimen. The analysis will report hazard ratios from a Cox proportional-hazards model.

IPD SHARING:
Plan to Share IPD: No
The data collected in this study are sensitive patient information. Due to privacy restrictions outlined in the informed consent form and institutional policies, the individual participant data will not be made publicly available.